CLINICAL TRIAL: NCT03974906
Title: Goal-directed Fluid Therapy in Elderly Patients Undergoing Lumbar Decompression Surgery in the Prone Position: A Randomized Controlled Clinical Trial
Brief Title: Goal-directed Fluid Therapy in Elderly Patients Undergoing Lumbar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Professor，Chairman, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PUMCH-GDT2
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Lactate Blood Increase; Fluid Overload; Postoperative Complications
Keywords: goal-directed fluid therapy; lactate acid level; postoperative complications; elderly patient; prone position; intraoperative hemodynamics
MeSH Terms: conditions — Hyperlactatemia; Edema; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients were assigned to one of the two groups (control group and GDT group) using a computer-generated randomization scheme.Allocation concealment was obtained using number labeled opaque envelopes that were opened just before the surgery. Data were collected by persons unaware of treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDT group (Experimental): The fluid in GDT group (Goal-directed fluid therapy) will be administered based upon real-time monitoring stroke volume variation and cardiac output achieved by the LiDCO monitoring system.
  Interventions: Other: Applying goal-directed fluid therapy by continuous hemodynamic monitoring system (LiDCO）
- Control group (No Intervention): Patients in the control group received conventional fluid therapy, decided by the attending anesthesiologists based on the patient's hemodynamic condition and responses, to maintain MAP >65 mm Hg, heart rate 50-100 bpm, and urine output >0.5 ml/kg/h.

INTERVENTIONS:
Other: Applying goal-directed fluid therapy by continuous hemodynamic monitoring system (LiDCO） — Applying continuous hemodynamic monitoring system ( LiDCO) to monitor Stroke Volume Variation and Cardiac Output and further manage intra-operative fluid therapy.
  Arms: GDT group

SUMMARY:
This is a randomized controlled clinical trial which investigates whether goal directed fluid therapy( GDT ) would show the evidence of benefit from GDT in terms of lactate kinetics then may reduce postoperative complications in patients undergoing spine surgery, especially in prone positions.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled clinical trial. Patients aged > 60 undergoing lumbar decompression surgery will be randomly assigned to either a GDT ( goal directed fluid therapy) group or a control group, who received conventional anesthesiologist-directed fluid therapy. Perioperative lactic acid concentrations with 7 different time point, intraoperative fluid balance and postoperative complications from admittance to 30 days after surgery were recorded. This RCT is conducted to show the evidence of benefit from GDT in terms of lactate kinetics then may reduce postoperative complications in patients undergoing spine surgery, especially in prone positions.

ELIGIBILITY:
Inclusion Criteria:

* age > 60 years, American Society of Anesthesiologists score II-III, and expected duration of operation > 2 h

Exclusion Criteria:

* Patients with severe cardiac arrhythmia (which would affect the accuracy of stroke volume variation as an indicator of fluid responsiveness), vascular disease (which would prohibit radial artery cannulation), and mental disorder were excluded

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Lactic acid concentrations throughout the perioperative | from 24 hours before surgery to 24 hours after the surgery
  the change of lactic acid concentrations(mmol/l) throughout the perioperative period

SECONDARY OUTCOMES:
intraoperative fluid balance, DO2I and predefined moderate or major postoperative complications in 30-day. | 30 days after the surgery
  Intraoperative fluid balance include the volumes of crystalloids(ml), colloids(ml) and total volumes of intravenous fluids and output of the patients during surgery.
  Derived DO2I(oxygen delivery index, ml/min·m2) variables were calculated according to standard formulae. The incidence of complications related to surgeries 30 days postoperatively. The complications include pneumonia, pulmonary embolism, cardiovascular events (myocardial infarction, heart failure), wound infection, gastrointestinal bleeding,nausea and vomitting，postoperative hemorrhage, ileus, deep venous thrombosis, cerebral infarction, cerebral embolism, cerebral hemorrhage, renal insufficiency and failure. Those complications are defined strictly to the reference published in 2009 New England Journal of Medicine （N Engl J Med. 2009 Oct 1;361:1368-75）

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishimoto Y, Yoshimura N, Muraki S, Yamada H, Nagata K, Hashizume H, Takiguchi N, Minamide A, Oka H, Kawaguchi H, Nakamura K, Akune T, Yoshida M. Associations between radiographic lumbar spinal stenosis and clinical symptoms in the general population: the Wakayama Spine Study. Osteoarthritis Cartilage. 2013 Jun;21(6):783-8. doi: 10.1016/j.joca.2013.02.656. Epub 2013 Mar 5. PMID 23473979
- [Background] Imajo Y, Taguchi T, Neo M, Otani K, Ogata T, Ozawa H, Miyakoshi N, Murakami H, Iguchi T. Complications of spinal surgery for elderly patients with lumbar spinal stenosis in a super-aging country: An analysis of 8033 patients. J Orthop Sci. 2017 Jan;22(1):10-15. doi: 10.1016/j.jos.2016.08.014. Epub 2016 Sep 16. PMID 27646205
- [Background] Li P, Qu LP, Qi D, Shen B, Wang YM, Xu JR, Jiang WH, Zhang H, Ding XQ, Teng J. Significance of perioperative goal-directed hemodynamic approach in preventing postoperative complications in patients after cardiac surgery: a meta-analysis and systematic review. Ann Med. 2017 Jun;49(4):343-351. doi: 10.1080/07853890.2016.1271956. Epub 2017 Feb 2. PMID 27936959
- [Background] Yuan J, Sun Y, Pan C, Li T. Goal-directed fluid therapy for reducing risk of surgical site infections following abdominal surgery - A systematic review and meta-analysis of randomized controlled trials. Int J Surg. 2017 Mar;39:74-87. doi: 10.1016/j.ijsu.2017.01.081. Epub 2017 Jan 23. PMID 28126672
- [Background] Bacchin MR, Ceria CM, Giannone S, Ghisi D, Stagni G, Greggi T, Bonarelli S. Goal-Directed Fluid Therapy Based on Stroke Volume Variation in Patients Undergoing Major Spine Surgery in the Prone Position: A Cohort Study. Spine (Phila Pa 1976). 2016 Sep 15;41(18):E1131-E1137. doi: 10.1097/BRS.0000000000001601. PMID 27046635
- [Background] Okorie ON, Dellinger P. Lactate: biomarker and potential therapeutic target. Crit Care Clin. 2011 Apr;27(2):299-326. doi: 10.1016/j.ccc.2010.12.013. PMID 21440203
- [Background] Myles PS, Bellomo R. Restrictive or Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Sep 27;379(13):1283. doi: 10.1056/NEJMc1810465. No abstract available. PMID 30257158
- [Result] Machado GC, Ferreira PH, Yoo RI, Harris IA, Pinheiro MB, Koes BW, van Tulder MW, Rzewuska M, Maher CG, Ferreira ML. Surgical options for lumbar spinal stenosis. Cochrane Database Syst Rev. 2016 Nov 1;11(11):CD012421. doi: 10.1002/14651858.CD012421. PMID 27801521